CLINICAL TRIAL: NCT00095147
Title: A Phase IIIB, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Comparative Study of Abatacept or Infliximab in Combination With Methotrexate in Controlling Disease Activity in Subjects With Rheumatoid Arthritis Having an Inadequate Clinical Response to Methotrexate
Brief Title: Abatacept and Infliximab in Combination With Methotrexate in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM101-043
Record Dates: First submitted 2004-11-01; First posted 2004-11-02 (Estimated); Results first posted 2011-01-21 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Methotrexate; Double-Blind Method; Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Abatacept (ABA) + Methotrexate (MTX) (double-blind [DB]) (Active Comparator): Days 1-365
  Interventions: Drug: Abatacept (ABA) + Methotrexate (MTX), double-blind (DB)
- Infliximab + MTX (DB) (Active Comparator): Days 1-365
  Interventions: Drug: Infliximab (INF) + MTX, DB
- Placebo + MTX (DB) (Placebo Comparator): Days 1-197
  Interventions: Drug: Placebo (PLA) + MTX, DB
- Placebo + MTX switched to abatacept + MTX (DB) (Experimental): Participants received placebo plus methotrexate for days 1-197, and abatacept plus methotrexate for days 198-365
  Interventions: Drug: PLA + MTX switched to ABA+ MTX, DB
- Abatacept (open-label) (Experimental): Days 365 to 729 All participants receive Active Drug
  Interventions: Drug: ABA, open-label (OL)

INTERVENTIONS:
Drug: Abatacept (ABA) + Methotrexate (MTX), double-blind (DB) — Abatacept, intravenous (IV) Solution, Infusion, Depends on participant weight, Monthly, 12 months.
  Other Names: Orencia
  Arms: Abatacept (ABA) + Methotrexate (MTX) (double-blind [DB])
Drug: Infliximab (INF) + MTX, DB — Infliximab, IV Solution, Infusion, Depends on participant weight, Every 2 Months, 12 months.
  Arms: Infliximab + MTX (DB)
Drug: Placebo (PLA) + MTX, DB — Placebo, IV Solution, Infusion, Depends on participant weight, Monthly, 6 months.
  Arms: Placebo + MTX (DB)
Drug: PLA + MTX switched to ABA+ MTX, DB — Placebo=IV Solution, Infusion, Depends on participant weight, Monthly, 6 months. Abatacept=IV Solution, Infusion, Depends on participant weight, Monthly, 6 months
  Other Names: Orencia
  Arms: Placebo + MTX switched to abatacept + MTX (DB)
Drug: ABA, open-label (OL) — Abatacept, IV solution, Infusion. Depends on participant weight, Monthly, 12+ months
  Other Names: Orencia
  Arms: Abatacept (open-label)

SUMMARY:
The purpose of this clinical research study is to learn if Abatacept or Infliximab in combination with Methotrexate demonstrate a greater reduction in disease activity over placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis
* At least 3 months prior treatment with Methotrexate (MTX)
* At least 10 swollen joints and 12 tender joints and C-Reactive Protein of at least 1 mg/dl
* Washout required for other disease modifying anti-rheumatic drugs (DMARDS)

Exclusion Criteria:

* participants who have failed more than 3 DMARDs
* participants previously treated with an approved biologic drug
* History of cancer in the last 5 years
* Severe or recurrent bacterial infection
* Any previous or current medical conditions that are contraindications to the use of TNF blocking agents
* Women of Child Bearing Potential

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2005-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (76):
- United States (19):
  - Local Institution, Huntsville, Alabama
  - Local Institution, Denver, Colorado
  - Local Institution, Boca Raton, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Largo, Florida
  - Local Institution, Indianapolis, Indiana
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Worcester, Massachusetts
  - Local Institution, Flowood, Mississippi
  - Local Institution, Syracuse, New York
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Bethlehem, Pennsylvania
  - Local Institution, Willow Grove, Pennsylvania
  - Local Institution, Austin, Texas
  - Local Institution, Dallas, Texas
- Argentina (5):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Quilmes, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, San Miguel de Tucumán, Tucumán Province
- Australia (7):
  - Local Institution, Cairns, Queensland
  - Local Institution, Cotton Tree, Queensland
  - Local Institution, Clayton, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Malvern, Victoria
  - Local Institution, Parkville, Victoria
  - Local Institution, Perth, Western Australia
- Brazil (5):
  - Local Institution, Curitiba, Paraná
  - Local Institution, Recife, Pernambuco
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, São Paulo, São Paulo
- Canada (11):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Hamilton, Ontario
  - Local Institution, Kitchener, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Ste-Foy, Quebec
  - Local Institution, Saskatoon, Saskatchewan
  - Local Institution, Kitchener
- Local Institution, Prague, Czechia
- Local Institution, Copenhagen, Denmark
- Mexico (6):
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, León, Guanajuato
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, San Luis Potosí City, San Luis Potosí
- Local Institution, Lima, Peru
- Poland (3):
  - Local Institution, Poznan
  - Local Institution, Sopot
  - Local Institution, Warsaw
- Local Institution, Rio Piedras, Puerto Rico
- Local Institution, Moscow, Russia
- South Africa (3):
  - Local Institution, Muckleneuk, Gauteng
  - Local Institution, Berea, KwaZulu-Natal
  - Local Institution, Panorama, Western Cape
- Local Institution, Seoul, South Korea
- Spain (4):
  - Local Institution, A Coruña
  - Local Institution, Barcelona
  - Local Institution, Córdoba
  - Local Institution, Madrid
- Sweden (5):
  - Local Institution, Falun
  - Local Institution, Linköping
  - Local Institution, Lund
  - Local Institution, Stockholm
  - Local Institution, Uppsala
- Switzerland (2):
  - Local Institution, Bern
  - Local Institution, Sankt Gallen

REFERENCES:
- [Derived] Schiff M, Keiserman M, Codding C, Songcharoen S, Berman A, Nayiager S, Saldate C, Li T, Aranda R, Becker JC, Lin C, Cornet PL, Dougados M. Efficacy and safety of abatacept or infliximab vs placebo in ATTEST: a phase III, multi-centre, randomised, double-blind, placebo-controlled study in patients with rheumatoid arthritis and an inadequate response to methotrexate. Ann Rheum Dis. 2008 Aug;67(8):1096-103. doi: 10.1136/ard.2007.080002. Epub 2007 Nov 29. PMID 18055472

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 748 participants enrolled in this study; 317 participants were not randomized or treated. 384 participants completed the double-blind period; 12 participants did not enter the open-label period.
Groups:
- Abatacept (ABA) + Methotrexate (MTX) [Double-blind (DB)]: Abatacept was administered intravenously (IV) on Days 1, 15, 29 and every 28 days thereafter for a total of 14 doses. Administration was as follows: 500 mg for participants < 60 kg, 750 mg for participants 60 to 100 kg and 1 gram for participants > 100 kg. All participants received a stable dose of MTX (minimum 15 mg weekly).
- Infliximab (INF) + MTX [DB]: Infliximab was given 3 mg/kg IV (approved labeled dose) on Days 1, 15, 43, 85 and every 56 days thereafter for a total of 8 doses. All participants received a stable dose of MTX (minimum 15 mg weekly)
- Placebo (PLA) + MTX [DB]: Normal saline was administered as placebo. All participants received a stable dose of MTX (minimum 15 mg weekly)
- PLA Switched to ABA + MTX [DB]: Normal saline was administered as placebo. All participants received a stable dose of MTX (minimum 15 mg weekly). After placebo treatment from Day 1-197, participants were reallocated to receive abatacept (weight based) plus a stable dose of MTX (minimum 15 mg weekly).
- ABA + MTX [Open-label (OL)]: All participants received ABA at a weight-tiered dose of 10 mg/kg plus a stable dose of MTX (minimum 15 mg weekly).
Period: Double-blind Period 1 (Days 1-197)
Arm/Group | Abatacept (ABA) + Methotrexate (MTX) [Double-blind (DB)] | Infliximab (INF) + MTX [DB] | Placebo (PLA) + MTX [DB] | PLA Switched to ABA + MTX [DB] | ABA + MTX [Open-label (OL)]
Started | 156 | 165 | 110 | 0 | 0
Completed | 147 | 152 | 107 | 0 | 0
Not Completed | 9 | 13 | 3 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 8 | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0 | 0 | 0
Not completed — Withdrawal of consent | 1 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 1 | 1 | 0 | 0 | 0
Period: Double-blind Period 2 (Days 198-365)
Arm/Group | Abatacept (ABA) + Methotrexate (MTX) [Double-blind (DB)] | Infliximab (INF) + MTX [DB] | Placebo (PLA) + MTX [DB] | PLA Switched to ABA + MTX [DB] | ABA + MTX [Open-label (OL)]
Started | 147 | 152 | 0 | 107 | 0
Completed | 139 | 141 | 0 | 104 | 0
Not Completed | 8 | 11 | 0 | 3 | 0
Not completed — Death | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 2 | 4 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 4 | 0 | 1 | 0
Not completed — Withdrawal of consent | 3 | 2 | 0 | 0 | 0
Not completed — Participant relocation | 1 | 0 | 0 | 1 | 0
Period: Long-term Extension Period
Arm/Group | Abatacept (ABA) + Methotrexate (MTX) [Double-blind (DB)] | Infliximab (INF) + MTX [DB] | Placebo (PLA) + MTX [DB] | PLA Switched to ABA + MTX [DB] | ABA + MTX [Open-label (OL)]
Started | 0 | 0 | 0 | 0 | 372
Completed | 0 | 0 | 0 | 0 | 327
Not Completed | 0 | 0 | 0 | 0 | 45
Not completed — Death | 0 | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 11
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 9
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 6
Not completed — Withdrawal of consent | 0 | 0 | 0 | 0 | 12
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1
Not completed — No longer meets study criteria | 0 | 0 | 0 | 0 | 1
Not completed — Participant chose to use Revellex | 0 | 0 | 0 | 0 | 1
Not completed — Leaving country | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- ABA + MTX [DB]: Abatacept was administered intravenously (IV) on Days 1, 15, 29 and every 28 days thereafter for a total of 14 doses. Administration was as follows: 500 mg for participants < 60 kg, 750 mg for participants 60 to 100 kg and 1 gram for participants > 100 kg. All participants received a stable dose of MTX (minimum 15 mg weekly).
- INF + MTX [DB]: Infliximab was given 3 mg/kg IV (approved labeled dose) on Days 1, 15, 43, 85 and every 56 days thereafter for a total of 8 doses. All participants received a stable dose of MTX (minimum 15 mg weekly)
- PLA + MTX [DB]: Normal saline was administered as placebo. All participants received a stable dose of MTX (minimum 15 mg weekly)
- Total: Total of all reporting groups
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB] | Total
Number analyzed (Participants) | 156 | 165 | 110 | 431
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (12.5) | 49.1 (12.0) | 49.4 (11.5) | 49.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 136 | 96 | 362
  Male | 26 | 29 | 14 | 69
Baseline Disease Activity Score (DAS) 28 (Erythrocyte Sedimentation Rate [ESR]) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or C-reactive protein (CRP), and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). A clinically significant response= decrease in DAS28 score of >1.2 from baseline.
  units on a scale | 6.9 (1.0) | 6.8 (0.9) | 6.8 (1.0) | 6.8 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: DB; Adjusted Mean Change From Baseline to Day 197 in Disease Activity Score (DAS) 28 Score (Erythrocyte Sedimentation Rate [ESR]) For ABA Versus PLA (Last Observation Carried Forward [LOCF] Analysis)
Description: The DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or C-reactive protein (CRP), and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). A clinically significant response is a decrease in DAS28 score of >1.2 from baseline.
Time Frame: Baseline (Day 1), 6 months (Day 197)
Population: The Intent-to-Treat (ITT) analysis population was defined to include all participants randomized into the study who received study medication. Participants were grouped according to the treatment or treatment regimen to which they were randomized. All participants who were randomized but never received study medication were excluded.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ABA + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 150 | 102
units on a scale | -2.53 (0.12) | -1.48 (0.15)
Statistical Analysis 1: Comparison: ABA + MTX [DB] vs PLA + MTX [DB]; The primary analysis was the comparison of abatacept versus placebo for changes from baseline to 6 months (Day 197) in the DAS28. This comparison was done using an analysis of covariance (ANCOVA) model with treatment group as the effect and baseline value as the covariate. A 95% confidence interval was computed for the treatment difference within the framework of the ANCOVA model; Test type: Superiority or Other; p < 0.001, ANCOVA; adjusted mean change from baseline = -1.04, 95% CI 2-sided [-1.42 to -0.67]

2. Secondary Outcome: DB; Adjusted Mean Change From Baseline to Day 197 in DAS 28 Score (ESR) For INF Versus PLA (LOCF Analysis)
Description: The DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or CRP, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). A clinically significant response is a decrease in DAS28 score of >1.2 from baseline.
Time Frame: Baseline (Day 1), 6 months (Day 197)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 156 | 102
units on a scale | -2.25 (0.12) | -1.48 (0.15)
Statistical Analysis 1: Comparison: INF + MTX [DB] vs PLA + MTX [DB]; Infliximab versus placebo were compared for changes from baseline to 6 months (Day 197) in the DAS28. This comparison was done using an analysis of covariance (ANCOVA) model with treatment group as the effect and baseline value as the covariate. A 95% confidence interval was computed for the treatment difference within the framework of the ANCOVA model; Test type: Superiority or Other; p < 0.001, ANCOVA; adjusted mean change from baseline = -0.77, 95% CI 2-sided [-1.14 to -0.39]

3. Secondary Outcome: DB; DAS 28 (ESR) Area Under The Curve (AUC) Over 12 Months For ABA Versus INF
Description: The DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or CRP, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). Clinically significant response= decrease in DAS28 score of >1.2 from baseline. DAS28 AUC can be calculated from the DAS28 score versus time curve, which provides an assessment of changes in disease activity over time.
Time Frame: From Day 1 through Day 365 (12 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ABA + MTX [DB[: Abatacept was administered intravenously (IV) on Days 1, 15, 29 and every 28 days thereafter for a total of 14 doses. Administration was as follows: 500 mg for participants < 60 kg, 750 mg for participants 60 to 100 kg and 1 gram for participants > 100 kg. All participants received a stable dose of MTX (minimum 15 mg weekly).
Arm/Group | ABA + MTX [DB[ | INF + MTX [DB]
Number analyzed (Participants) | 150 | 156
units on a scale | 1638.6 (395.81) | 1657.5 (460.52)

4. Secondary Outcome: DB; Percentage of Participants With Clinically Meaningful Health Assessment Questionnaire-Disability Index (HAQ-DI) Response at Day 197
Description: The disability section of the full HAQ includes 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. The questions are evaluated on a 4-point scale: 0=without any difficulty, 1= with some difficulty, 2= with much difficulty, and 3= unable to do. Higher scores= greater dysfunction. A disability index was calculated by summing the worst scores in each domain and dividing by the number of domains answered. Clinically meaningful HAQ response=an improvement of at least 0.3 units from baseline in HAQ disability Index.
Time Frame: DB Day 197
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 156 | 165 | 110
percentage of participants | 61.5 | 58.8 | 40.9
Statistical Analysis 1: Comparison: ABA + MTX [DB] vs PLA + MTX [DB]; Comparisons were made between ABA and PLA at Day 197 using a continuity corrected Chi-square test. All tests and confidence intervals for treatment comparison were two-sided; Test type: Superiority or Other; p = 0.001, Chi-squared, Corrected; Estimate of difference from placebo = 20.6, 95% CI 2-sided [7.7 to 33.6]
Statistical Analysis 2: Comparison: INF + MTX [DB] vs PLA + MTX [DB]; Comparisons were made between INF and PLA at Day 197 using a continuity corrected Chi-square test. All tests and confidence intervals for treatment comparison were two-sided; Test type: Superiority or Other; p = 0.005, Chi-squared, Corrected; Estimate of difference from placebo = 17.9, 95% CI 2-sided [5.1 to 30.7]

5. Secondary Outcome: DB; Percentage of Participants With Clinically Meaningful Health Assessment Questionnaire-Disability Index (HAQ-DI) Response at Day 365
Description: as for outcome 4
Time Frame: DB Day 365
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- PLA + MTX [DB]: Normal saline was administered as placebo. All participants received a stable dose of MTX (minimum 15 mg weekly). After placebo treatment from Day 1-197, participants were reallocated to receive abatacept (weight based) plus a stable dose of MTX (minimum 15 mg weekly).
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 156 | 165 | 110
percentage of participants | 57.7 | 52.7 | 57.3

6. Secondary Outcome: DB; Adjusted Mean Change From Baseline to Day 197 in HAQ-DI (LOCF Analysis)
Description: as for outcome 4
Time Frame: Baseline (Day 1), 6 months (Day 197)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 156 | 164 | 109
units on a scale
  HAQ-DI | -0.69 (0.05) | -0.61 (0.05) | -0.31 (0.06)
  HAQ-DI component: activities | -0.61 (0.06) | -0.54 (0.06) | -0.22 (0.08)
  HAQ-DI component: dressing and grooming | -0.69 (0.06) | -0.57 (0.06) | -0.37 (0.07)
  HAQ-DI component: eating | -0.79 (0.06) | -0.77 (0.06) | -0.36 (0.08)
  HAQ-DI component: grip | -0.73 (0.07) | -0.70 (0.07) | -0.26 (0.08)
  HAQ-DI component: hygiene | -0.64 (0.07) | -0.48 (0.07) | -0.26 (0.08)
  HAQ-DI component: reach | -0.72 (0.07) | -0.64 (0.07) | -0.30 (0.08)
  HAQ-DI component: arising | -0.70 (0.06) | -0.68 (0.06) | -0.39 (0.07)
  HAQ-DI component: walking | -0.58 (0.06) | -0.56 (0.06) | -0.23 (0.07)
Statistical Analysis 1: Comparison: ABA + MTX [DB] vs PLA + MTX [DB]; Adjusted mean change in HAQ-DI from baseline to 6 months (Day 197) was compared between ABA and PLA. This comparison was done using an analysis of covariance (ANCOVA) model with treatment group as the effect and baseline value as the covariate. A 95% confidence interval was computed for the treatment difference within the framework of the ANCOVA model; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference from placebo = -0.38, 95% CI 2-sided [-0.53 to -0.23]
Statistical Analysis 2: Comparison: INF + MTX [DB] vs PLA + MTX [DB]; Adjusted mean change in HAQ-DI from baseline to 6 months (Day 197) was compared between INF and PLA. This comparison was done using an analysis of covariance (ANCOVA) model with treatment group as the effect and baseline value as the covariate. A 95% confidence interval was computed for the treatment difference within the framework of the ANCOVA model; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference from placebo = -0.30, 95% CI 2-sided [-0.45 to -0.15]

7. Secondary Outcome: DB; Adjusted Mean Change From Baseline to Day 365 in HAQ-DI (LOCF Analysis)
Description: as for outcome 4
Time Frame: Baseline (Day 1), 12 months (Day 365)
Population: Intent-to-Treat (ITT) Population: all participants randomized into the study receiving study medication, grouped according to randomization treatment. All participants randomized but never receiving study medication excluded. Although 3 participants in PLA group discontinued before Day 197, 2 of these patients were included in the LOCF analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 156 | 164 | 109
units on a scale
  HAQ-DI | -0.67 (0.05) | -0.59 (0.05) | -0.56 (0.06)
  HAQ-DI component: activities | -0.55 (0.07) | -0.52 (0.07) | -0.55 (0.08)
  HAQ-DI component: dressing and grooming | -0.72 (0.06) | -0.60 (0.06) | -0.56 (0.07)
  HAQ-DI component: eating | -0.80 (0.06) | -0.73 (0.06) | -0.71 (0.08)
  HAQ-DI component: grip | -0.77 (0.07) | -0.64 (0.07) | -0.56 (0.08)
  HAQ-DI component: hygiene | -0.53 (0.07) | -0.45 (0.07) | -0.42 (0.09)
  HAQ-DI component: reach | -0.77 (0.07) | -0.66 (0.07) | -0.53 (0.08)
  HAQ-DI component: arising | -0.68 (0.06) | -0.64 (0.06) | -0.61 (0.07)
  HAQ-DI component: walking | -0.54 (0.06) | -0.55 (0.06) | -0.47 (0.07)

8. Secondary Outcome: DB; Adjusted Mean Change From Baseline to Day 197 in SF-36 Physical Component Summary (PCS) and Mental Component Summary (MCS)
Description: The SF-36 is a validated instrument measuring health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores (1) physical component summary=physical functioning, role-physical, bodily pain, and general health; (2) mental component summary=vitality, social functioning, role-emotional, and mental health. There is no total overall score; scoring is done for both subscores and summary scores. For subscores and summary scores, 0 =worst score (or quality of life) and 100=best score. Change from Baseline= post-Baseline - Baseline value.
Time Frame: Baseline (Day 1), 6 months (Day 197)
Population: ITT population, all participants randomized into the study receiving study medication. Participants grouped according to the treatment to which they were randomized. All randomized participants who never received study medication were excluded. SF-36 component scores were not presented in tabular form.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 154 | 163 | 109
units on a scale
  SF-36 Physical Component Summary | 8.36 (0.69) | 7.66 (0.67) | 4.34 (0.82)
  SF-36 Mental Component Summary | 5.14 (0.79) | 4.32 (0.76) | 1.64 (0.93)
Statistical Analysis 1: Comparison: ABA + MTX [DB] vs PLA + MTX [DB]; Adjusted mean change in SF-36 physical component summary from baseline to 6 months (Day 197) was compared between ABA and PLA. This comparison was done using an analysis of covariance (ANCOVA) model with treatment group as the effect and baseline value as the covariate. A 95% confidence interval was computed for the treatment difference within the framework of the ANCOVA model; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference from placebo (PCS) = 4.02, 95% CI 2-sided [1.92 to 6.12]
Statistical Analysis 2: Comparison: ABA + MTX [DB] vs PLA + MTX [DB]; Adjusted mean change in SF-36 mental component summary from baseline to 6 months (Day 197) was compared between ABA and PLA. This comparison was done using an analysis of covariance (ANCOVA) model with treatment group as the effect and baseline value as the covariate. A 95% confidence interval was computed for the treatment difference within the framework of the ANCOVA model; Test type: Superiority or Other; p = 0.004, ANCOVA; Difference from placebo (MCS) = 3.51, 95% CI 2-sided [1.10 to 5.91]
Statistical Analysis 3: Comparison: INF + MTX [DB] vs PLA + MTX [DB]; Adjusted mean change in SF-36 physical component summary from baseline to 6 months (Day 197) was compared between INF and PLA. This comparison was done using an analysis of covariance (ANCOVA) model with treatment group as the effect and baseline value as the covariate. A 95% confidence interval was computed for the treatment difference within the framework of the ANCOVA model; Test type: Superiority or Other; p = 0.002, ANCOVA; Difference from placebo (PCS) = 3.32, 95% CI 2-sided [1.25 to 5.40]
Statistical Analysis 4: Comparison: INF + MTX [DB] vs PLA + MTX [DB]; Adjusted mean change in SF-36 mental component summary from baseline to 6 months (Day 197) was compared between INF and PLA. This comparison was done using an analysis of covariance (ANCOVA) model with treatment group as the effect and baseline value as the covariate. A 95% confidence interval was computed for the treatment difference within the framework of the ANCOVA model; Test type: Superiority or Other; p = 0.027, ANCOVA; Difference from placebo (MCS) = 2.68, 95% CI 2-sided [0.31 to 5.05]

9. Secondary Outcome: DB; Adjusted Mean Change From Baseline to Day 365 in SF-36 Physical Component Summary (PCS) and Mental Component Summary (MCS)
Description: as for outcome 8
Time Frame: Baseline (Day 1), 12 months (Day 365)
Population: ITT Population: all participants randomized into the study receiving study medication, grouped according to randomization treatment. Although 3 participants in PLA group discontinued before Day 197, 2 of these patients were included in the LOCF analysis. SF-36 component scores were not presented in tabular form.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 154 | 163 | 109
units on a scale
  SF-36 Physical Component Summary | 9.52 (0.70) | 7.59 (0.68) | 8.00 (0.83)
  SF-36 Mental Component Summary | 5.96 (0.81) | 4.03 (0.79) | 5.85 (0.97)

10. Secondary Outcome: DB; Percentage of Participants With Good, Moderate, or No Response According to European League Against Rheumatism (EULAR) at Day 365
Description: The DAS28 is a continuous disease measure composite of 4 variables: 28 tender joint count, 28 swollen joint count, ESR or CRP, and participant assessment of disease activity measure on a visual analogue scale. High disease activity= > 5.1, low disease activity= < 3.2, and remission= < 2.6. Clinically significant response= decrease of >1.2 from baseline. Utilizing EULAR response criteria, DAS28 categorical responses define a good (absolute: <3.2 or >1.2 improvement from baseline [BL]), moderate (absolute: 3.2-5.1 or 0.6-1.2 change from BL), or no response (absolute: >5.1 or <0.6 change from BL)
Time Frame: DB Day 365
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 150 | 157 | 102
percentage of participants
  No response | 27.3 | 36.3 | 23.5
  Moderate response | 40.7 | 45.2 | 49.0
  Good response | 32.0 | 18.5 | 27.5

11. Secondary Outcome: DB; Percentage of Participants With American College of Rheumatology (ACR) Responses at Day 197
Description: The ACR 20 definition of improvement is a 20% improvement from baseline in the number of tender and swollen joint counts, and a 20% improvement from baseline in 3 of the remaining 5 core set measures: participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function and acute phase reactant value (C-reactive protein [CRP]). The evaluation for 50% improvement (ACR 50) and 70% improvement (ACR 70) follow similarly.
Time Frame: DB Day 197
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 156 | 165 | 110
percentage of participants
  Day 197, ACR 20 | 66.7 | 59.4 | 41.8
  Day 197, ACR 50 | 40.4 | 37.0 | 20.0
  Day 197, ACR 70 | 20.5 | 24.2 | 9.1

12. Secondary Outcome: DB; Percentage of Participants With American College of Rheumatology (ACR) Responses at Day 365
Description: as for outcome 11
Time Frame: DB Day 365
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 156 | 165 | 110
percentage of participants
  Day 365, ACR 20 | 72.4 | 55.8 | 68.2
  Day 365, ACR 50 | 45.5 | 36.4 | 50.9
  Day 365, ACR 70 | 26.3 | 20.6 | 29.1

13. Secondary Outcome: DB; Number of Participants With Death, Serious Adverse Events (SAEs), Related SAEs, SAEs Leading to Discontinuation, AEs, Related AEs, and AEs Leading to Discontinuation From Day 1 Through Day 197
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event.
Time Frame: From Baseline (Day 1) through Day 197, and up to 56 days after last dose if occurring on-study
Population: The As-Treated analysis population contained all participants who received at least one dose of double-blind study medication, and participants were grouped on an as-assigned or randomized basis unless the participant received the incorrect medication for the entire period of treatment.
Measure: Number; unit: participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 156 | 165 | 110
participants
  Deaths | 1 | 1 | 0
  SAEs | 8 | 19 | 13
  Related SAEs | 3 | 8 | 3
  SAEs Leading to Discontinuation | 2 | 4 | 0
  AEs | 129 | 140 | 92
  Related AEs | 64 | 74 | 46
  AEs Leading to discontinuation | 3 | 8 | 1

14. Secondary Outcome: DB; Number of Participants With AEs of Special Interest From Day 1 Through Day 197
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. AEs of special interest are those AEs that may be associated with the use of immunomodulatory drugs, including all infections, serious infections, autoimmune disorders; malignancies; and acute infusional AEs (pre-specified AEs occurring within 1 hour of start of infusion).
Time Frame: From Baseline (Day 1) through Day 197, and up to 56 days after last dose if occurring on-study
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 156 | 165 | 110
participants
  Pre-specified infections | 12 | 18 | 8
  Neoplasms: Benign, malignant, and unspecified | 1 | 2 | 1
  Prespecified autoimmune symptoms and disorders | 1 | 1 | 1
  Pre-specified infusional AEs | 8 | 30 | 11

15. Secondary Outcome: DB; Number of Participants With Death, Serious Adverse Events (SAEs), Related SAEs, SAEs Leading to Discontinuation, AEs, Related AEs, and AEs Leading to Discontinuation From Day 1 Through Day 365
Description: as for outcome 13
Time Frame: From Baseline (Day 1) through Day 365, and up to 56 days after last dose if occurring on-study
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB]
Number analyzed (Participants) | 156 | 165
participants
  Deaths | 1 | 2
  SAEs | 15 | 30
  Related SAEs | 5 | 14
  SAEs Leading to Discontinuation | 4 | 6
  AEs | 139 | 154
  Related AEs | 72 | 96
  AEs Leading to discontinuation | 5 | 12

16. Secondary Outcome: DB; Number of Participants With Death, Serious Adverse Events (SAEs), Related SAEs, SAEs Leading to Discontinuation, AEs, Related AEs, and AEs Leading to Discontinuation From Day 198 Through Day 365 in Participants Receiving Placebo Switched to Abatacept
Description: as for outcome 13
Time Frame: From Day 198 through Day 365, and up to 56 days after last dose if occurring on-study
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | PLA Switched to ABA + MTX [DB]
Number analyzed (Participants) | 110
participants
  Deaths | 1
  SAEs | 12
  Related SAEs | 3
  SAEs Leading to Discontinuation | 0
  AEs | 71
  Related AEs | 26
  AEs Leading to discontinuation | 0

17. Primary Outcome: OL; Number of Participants With Death, Serious Adverse Events (SAEs), Related SAEs, SAEs Leading to Discontinuation, Adverse Events (AEs), Related AEs, and AEs Leading to Discontinuation
Description: as for outcome 13
Time Frame: From beginning of OL (Day 366) through end of OL (range from 1.9 months to 42.3 months)
Population: All Treated Population, all participants who entered the open-label period and received at least one dose of abatacept at any time during this period.
Measure: Number; unit: participants
Groups:
- ABA + MTX [OL]: All participants received ABA at a weight-tiered dose of 10 mg/kg plus a stable dose of MTX (minimum 15 mg weekly).
Arm/Group | ABA + MTX [OL]
Number analyzed (Participants) | 372
participants
  Deaths | 3
  SAEs | 90
  Related SAEs | 12
  SAEs Leading to Discontinuation | 5
  AEs | 349
  Related AEs | 165
  AEs Leading to discontinuation | 10

18. Primary Outcome: OL; Number of Participants With AEs of Special Interest
Description: as for outcome 14
Time Frame: From beginning of OL (Day 366) through end of OL (range from 1.9 months to 42.3 months)
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | ABA + MTX [OL]
Number analyzed (Participants) | 372
participants
  Infections | 277
  Malignant neoplasms | 3
  Benign and unspecified neoplasms | 18
  Prespecified autoimmune symptoms and disorders | 13
  Pre-specified peri-infusional AEs | 50
  Pre-specified acute infusional AEs | 28

19. Primary Outcome: OL; Number of Participants With Select Hematologic Laboratory Abnormalities
Description: High=greater than Upper Normal Limit (ULN), Low=lower than Lower Normal Limit (LLN). LLN/ULN= Hemoglobin (HGB): >3 g/dL decrease from Baseline (BL); Hematocrit: <0.75 x BL; Erythrocytes: <0.75 x BL; Platelets (PLT): <0.67 x LLN/>1.5 x ULN; Leukocytes: <0.75 x LLN/ >1.25 x ULN; neutrophils+bands: <1.0 x 10^3 c/uL; lymphocytes: <0.750 x 10^3 c/uL/ >7.50 x 10^3 c/uL; monocytes: >2000 mm3; eosinophils: >0.750 x 10^3 c/uL;
Time Frame: From Day 366 through end of OL (range from 1.9 months to 42.3 months)
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | ABA + MTX [OL]
Number analyzed (Participants) | 372
participants
  Low HGB (>3g/dL decrease from BL), n=372 | 9
  Low hematocrit (< 0.75 x BL), n=372 | 7
  Low erythrocytes (<0.75 x BL), n=372 | 6
  Low PLT (<0.67 x LLN), n=370 | 2
  High leukocytes (>1.25 x ULN), n=372 | 29
  Low neutrophils + bands (<1.0 x 10^3 c/uL), n=372 | 1
  Low lymphocytes (<0.75 x 10^3 c/uL), n=372 | 12
  High monocytes (>2000/mm^3), n=372 | 3
  High eosinophils (>0.750 x 10^3 c/uL), n=372 | 15

20. Primary Outcome: OL; Number of Participants With Select Blood Chemistry Laboratory Abnormalities
Description: Low=lower than LLN, High=greater than ULN. LLN/ULN= Alkaline phosphatase (ALP): >2 x ULN; aspartate aminotransferase (AST): >3 x ULN; alanine aminotransferase (ALT): >3 x ULN; G-Glutamyl transferase (GGT): >2 x ULN; Bilirubin: >2 x ULN; blood urea nitrogen (BUN): >2 x BL; creatinine: >4 x BL
Time Frame: From Day 366 through end of OL (range from 1.9 months to 42.3 months)
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | ABA + MTX [OL]
Number analyzed (Participants) | 371
participants
  High ALP (>2 x ULN) | 1
  High AST (>3 x ULN) | 4
  High ALT (>3 x ULN) | 11
  High GGT (>2 x ULN) | 16
  High total bilirubin (>2 x ULN) | 1
  High BUN (>2 x BL) | 17
  High creatinine (>1.5 increase from BL) | 44

21. Secondary Outcome: DB; Number of Participants With AEs of Special Interest From Day 1 Through Day 365
Description: as for outcome 14
Time Frame: From Baseline (Day 1) through Day 365, and up to 56 days after last dose if occurring on-study
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB]
Number analyzed (Participants) | 156 | 165
participants
  Pre-specified infections | 16 | 30
  Neoplasms:Benign, malignant, and unspecified | 1 | 2
  Prespecified autoimmune symptoms and disorders | 2 | 1
  Pre-specified infusional AEs | 11 | 41

22. Secondary Outcome: DB; Number of Participants With AEs of Special Interest From Day 198 Through Day 365 in Participants Receiving Placebo Switched to Abatacept
Description: as for outcome 14
Time Frame: From Day 198 through Day 365, and up to 56 days after last dose if occurring on-study
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | PLA Switched to ABA + MTX [DB]
Number analyzed (Participants) | 110
participants
  Pre-specified infections | 3
  Prespecified autoimmune symptoms and disorders | 1
  Pre-specified infusional AEs | 5

23. Secondary Outcome: DB; Number of Participants With Significant Changes in Mean Systolic and Diastolic Blood Pressure During Days 1 Through 197 and Days 1 Through 365
Description: Seated Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) were assessed as clinically significant or relevant at the discretion of the Clinical Investigator. Criteria may have varied between institutions.
Time Frame: From Baseline (Day 1) through Day 197, or Day 1 through Day 365, and up to 56 days after last dose if occurring on-study
Population: As-Treated Population
Measure: Number; unit: participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 156 | 165 | 110
participants
  Days 1-197 | 0 | 0 | 0
  Days 1-365 | 0 | 0 | 0

24. Secondary Outcome: DB; Number of Participants With Significant Changes in Mean Heart Rate During Days 1 Through 197 and Days 1 Through 365
Description: Heart Rate (HR) was assessed as clinically significant or relevant at the discretion of the Clinical Investigator. Criteria may have varied between institutions.
Time Frame: as for outcome 23
Population: As Treated Population.
Measure: Number; unit: participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 156 | 165 | 110
participants
  Days 1-197 | 0 | 0 | 0
  Days 1-365 | 0 | 0 | 0

25. Secondary Outcome: DB; Number of Participants With Significant Changes in Mean Temperature During Days 1 Through 197 and Days 1 Through 365
Description: Temperature (T) was assessed as clinically significant or relevant at the discretion of the Clinical Investigator. Criteria may have varied between institutions.
Time Frame: From Baseline (Day 1) through Day 197, and up to 56 days after last dose if occurring on-study
Population: As Treated Population.
Measure: Number; unit: participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 156 | 165 | 110
participants
  Days 1-197 | 0 | 0 | 0
  Days 1-365 | 0 | 0 | 0

26. Secondary Outcome: DB; Number of Participants With Select Hematologic and Blood Chemistry Laboratory Abnormalities on Days 1 Through 197
Description: High=greater than Upper Normal Limit (ULN), Low=lower than Lower Normal Limit (LLN). LLN/ULN= Hemoglobin (HGB): >3 g/dL decrease from Baseline (BL); Hematocrit: <0.75 x BL; Platelets (PLT): <0.67 x LLN/>1.5 x ULN; Leukocytes: <0.75 x LLN/ >1.25 x ULN; neutrophils+bands: <1.0 x 10^3 c/uL; aspartate aminotransferase (AST): >3 x ULN; alanine aminotransferase (ALT): >3 x ULN; creatinine: >4 x BL
Time Frame: From Baseline (Day 1) through Day 197, and up to 56 days after last dose if occurring on-study
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 155 | 162 | 108
participants
  Low HGB (n=155, n=162, n=108) | 1 | 1 | 1
  Low hematocrit (n=155, n=162, n=108) | 0 | 2 | 0
  Low PLT (n=154, n=160, n=108) | 1 | 2 | 0
  High PLT (n=154, n=160, n=108) | 0 | 0 | 1
  Low leukocytes (n=155, n=162, n=108) | 0 | 1 | 0
  High leukocytes (n=155, n=162, n=108) | 6 | 12 | 16
  Low neutrophils + bands (n=155, n=162, n=108) | 0 | 0 | 1
  High AST (n=155, n=162, n=108) | 3 | 3 | 1
  High ALT (n=155, n=162, n=108) | 3 | 2 | 3
  High creatinine (n=155, n=162, n=108) | 6 | 9 | 5

27. Secondary Outcome: DB; Number of Participants With Select Hematologic and Blood Chemistry Laboratory Abnormalities on Days 1 Through 365
Description: as for outcome 26
Time Frame: From Baseline (Day 1) through Day 365, and up to 56 days after last dose if occurring on-study
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA Switched to ABA + MTX [DB]
Number analyzed (Participants) | 156 | 164 | 109
participants
  Low HGB (n=156, n=164, n=109) | 2 | 1 | 1
  Low hematocrit (n=156, n=164, n=109) | 1 | 2 | 0
  Low PLT (n=155, n=162, n=109) | 1 | 2 | 0
  High PLT (n=155, n=162, n=109) | 0 | 0 | 1
  Low leukocytes (n=156, n=164, n=109) | 0 | 1 | 0
  High leukocytes (n=156, n=164, n=109) | 7 | 22 | 20
  Low neutrophils + bands (n=156, n=164, n=109) | 0 | 0 | 1
  High AST (n=156, n=164, n=109) | 4 | 6 | 3
  High ALT (n=156, n=164, n=109) | 3 | 7 | 5
  High creatinine (n=156, n=164, n=109) | 10 | 13 | 7

28. Secondary Outcome: DB; Number of Participants With Anti-Abatacept Antibodies From Day 1 Through Day 365 (Electrochemiluminescent [ECL] Immunoassay)
Description: ECL screened sera for drug-specific antibodies, immunocompetition was used to identify specific anti-Abatacept reactivity. Cytotoxic leukocyte antigen 4 (CTLA4) and Possibly Immunoglobulin (Ig) Category=reactivity against extracellular domain of human CTLA4, constant regions of human IgG1, or both (CTLA4Ig; Abatacept molecule). Ig and/or Junction Category=reactivity against constant regions and/or hinge region of human IgG1. Drug-induced seropositivity was defined as a post-baseline titer higher than Baseline, or any post-baseline positivity if Baseline value was missing.
Time Frame: Day 1 through day 365
Population: The immunogenicity analysis population included participants who received at least one dose of abatacept and had immunogenicity samples collected at baseline and at least one post-baseline treatment visit.
Measure: Number; unit: participants
Arm/Group | ABA + MTX [DB] | PLA Switched to ABA + MTX [DB]
Number analyzed (Participants) | 156 | 110
participants
  CTLA4 and Possibly Ig | 0 | 0
  Ig and/or Junction | 0 | 0

29. Secondary Outcome: DB; Percentage of Participants With Antibodies Against Infliximab (Human Anti-chimeric Antibody [HACA]) From Day 1 Through Day 365
Description: Infliximab levels were measured using a microplate enzyme-linked immunosorbant assay (ELISA) with infliximab bound to immobilized recombinant tumor necrosis factor (TNF)-alpha. Bound infliximab is detected utilizing a horseradish peroxidase-conjugated anti-human IgG Fc(fragment, crystallizable region)-specific). The enzyme turns over the substrate O-phenlenediamine to a chromogenic product that is measured at 490 nm. The cut-off value was 1.40 ug/mL; this was based on the mean (+ 3 SD) value in serum samples from 40 participants who had never received infliximab.
Time Frame: Day 1 through day 365
Population: The immunogenicity analysis population included participants who received at least one dose of infliximab and had immunogenicity samples collected at baseline and at least one post-baseline treatment visit.
Measure: Number; unit: percentage of participants
Arm/Group | INF + MTX [DB]
Number analyzed (Participants) | 163
percentage of participants
  Overall anti-HACA | 62.0
  Overall indeterminate anti-HACA | 73.0
  Day 1 anti-HACA | 0
  Day 1 indeterminate anti-HACA | 3.7
  Day 113 anti-HACA | 20.0
  Day 113 indeterminate anti-HACA | 74.7
  Day 197 anti-HACA | 42.2
  Day 197 indeterminate anti-HACA | 33.3
  Day 309 anti-HACA | 53.6
  Day 309 indeterminate anti-HACA | 29.7
  Post Day 28 anti-HACA | 52.2
  Post Day 28 indeterminate anti-HACA | 27.5
  Discontinued, overall anti-HACA | 60.9
  Discontinued, overall indeterminate anti-HACA | 47.8
  Discontinued, post day 28 anti-HACA | 55.0
  Discontinued, post day 28 indeterminate anti-HACA | 25.0
  Discontinued, post day 56 anti-HACA | 72.7
  Discontinued, post day 56 indeterminate anti-HACA | 9.1
  Discontinued, post day 85 anti-HACA | 88.9
  Discontinued, post day 85 indeterminate anti-HACA | 0
  Missed doses, overall anti-HACA | 73.1
  Missed doses, overall indeterminate anti-HACA | 76.9
  Missed 1 dose, anti-HACA | 72.0
  Missed 1 dose, indeterminate anti-HACA | 76.0
  Missed >1 dose, anti-HACA | 100.0
  Missed >1 dose, indeterminate anti-HACA | 100.0

30. Primary Outcome: OL; Mean Change From Baseline to Day 365 in Hemoglobin, Total Protein, and Albumin
Description: Hemoglobin (HGB): >3 g/dL decrease from BL; total protein: < 0.9 x LLN, >1.1 x ULN; albumin:<0.9 x LLN
Time Frame: Baseline (Day 1), Day 365
Population: Number of Participants Analyzed=All Treated Population, all participants who entered the open-label period and received at least one dose of abatacept at any time during this period. Treatment groups represent treatment received in the DB period. n=number of participants with data available.
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 131 | 136 | 104
g/dL
  HGB (n=131, n=135, n=103) | 0.53 (0.09) | 0.24 (0.09) | 0.43 (0.09)
  Total protein (n=131, n=136, n=104) | -0.09 (0.04) | 0.11 (0.04) | -0.12 (0.04)
  Albumin (n=131, n=136, n=104) | 0.12 (0.03) | 0.00 (0.03) | 0.05 (0.03)

31. Primary Outcome: OL; Mean Change From Baseline to Day 365 in Platelets
Description: Platelets (PLT): <0.67 x LLN, >1.5 x ULN
Time Frame: Baseline (Day 1), Day 365
Population: as for outcome 30
Measure: Mean (Standard Error); unit: 10^9 c/L
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 129 | 129 | 102
10^9 c/L | -42.4 (5.20) | -35.5 (6.93) | -28.4 (6.75)

32. Primary Outcome: OL; Mean Change From Baseline to Day 365 in Hematocrit
Description: Hematocrit: <0.75 x BL
Time Frame: Baseline (Day 1), Day 365
Population: as for outcome 30
Measure: Mean (Standard Error); unit: percentage red blood cells
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 129 | 134 | 102
percentage red blood cells | 1.44 (0.29) | 0.51 (0.27) | 1.03 (0.27)

33. Primary Outcome: OL; Mean Change From Baseline to Day 365 in White Blood Cells
Description: Leukocytes: <0.75 x LLN, >1.25 x ULN; neutrophils+bands: <1.0 x 10^3 c/uL; eosinophils: >0.750 x 10^3 c/uL; basophils: > 400 mm3; monocytes: >2000 mm3; lymphocytes: <0.750 x 10^3 c/uL, >7.50 x 10^3 c/uL.
Time Frame: Baseline (Day 1), Day 365
Population: as for outcome 30
Measure: Mean (Standard Error); unit: 10^3 c/uL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 131 | 134 | 104
10^3 c/uL
  Leukocytes (n=131, n=134, n=103) | -0.95 (0.23) | -0.90 (0.21) | -0.84 (0.23)
  Neutrophils + bands (n=130, n=130, n=104) | -0.91 (0.20) | -1.14 (0.20) | -1.05 (0.22)
  Basophils (n=130, n=130, n=101) | -0.01 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Monocytes (n=130, n=130, n=101) | -0.01 (0.02) | -0.01 (0.02) | 0.02 (0.02)
  Eosinophils (n=130, n=130, n=101) | -0.04 (0.01) | -0.02 (0.02) | -0.03 (0.01)
  Lymphocytes (n=130, n=130, n=101) | 0.03 (0.07) | 0.24 (0.06) | 0.22 (0.08)

34. Primary Outcome: OL; Mean Change From Baseline to Day 365 in Erythrocytes
Description: Erythrocytes: <0.75 x BL
Time Frame: Baseline (Day 1), Day 365
Population: as for outcome 30
Measure: Mean (Standard Error); unit: 10^6 c/uL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 131 | 135 | 103
10^6 c/uL | 0.09 (0.03) | 0.00 (0.03) | 0.006 (0.03)

35. Primary Outcome: OL; Mean Change From Baseline to Day 365 in Electrolytes
Description: Sodium (Na): <0.95 x LLN, >1.05 x ULN; potassium (K): <0.9 x LLN, >1.1 x ULN; chloride (Cl): <0.9 x LLN, >1.1 x ULN
Time Frame: Baseline (Day 1), Day 365
Population: as for outcome 30
Measure: Mean (Standard Error); unit: mEq/L
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 131 | 136 | 104
mEq/L
  Na (n=131, n=136, n=104) | -1.62 (0.29) | -1.57 (0.33) | -1.09 (0.38)
  K (n=131, n=135, n=104) | -0.03 (0.04) | -0.07 (0.04) | -0.03 (0.05)
  Cl (n=131, n=136, n=104) | -1.40 (0.28) | -1.18 (0.31) | -1.06 (0.33)

36. Primary Outcome: OL; Mean Change From Baseline to Day 365 in Bilirubin, Blood Urea Nitrogen, Creatinine, Calcium, Phosphorous, Serum Glucose, Fasting Serum Glucose, and Uric Acid
Description: Bilirubin: >2 x ULN; blood urea nitrogen (BUN): >2 x BL; creatinine: >4 x BL; calcium (Ca): <0.8 x LLN, >1.2 x ULN; phosphorous (P): <0.75 x LLN, >1.2 5 x ULN; serum glucose (Glu): <65 mg/dL, >220 mg/dL; fasting serum Glu: <0.8 x LLN, >1.5 x ULN; uric acid: >1.5 x ULN;
Time Frame: Baseline (Day 1), Day 365
Population: as for outcome 30
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 131 | 136 | 104
mg/dL
  Creatinine (n=131, n=136, n=104) | 0.03 (0.02) | 0.02 (0.01) | 0.01 (0.02)
  BUN (n=131, n=136, n=104) | -0.31 (0.41) | -0.52 (0.40) | 0.10 (0.53)
  Ca (n=131, n=136, n=104) | 0.14 (0.04) | 0.08 (0.03) | 0.14 (0.04)
  P (n=131, n=136, n=104) | 0.03 (0.05) | -0.01 (0.05) | 0.05 (0.05)
  Uric Acid (n=131, n=136, n=104) | 0.09 (0.08) | 0.08 (0.10) | 0.04 (0.12)
  Total bilirubin (n=131, n=134, n=104) | 0.06 (0.01) | 0.04 (0.02) | 0.03 (0.02)
  Serum glucose (n=131, n=136, n=104) | 5.66 (2.41) | 2.49 (3.15) | 3.03 (2.16)

37. Primary Outcome: OL; Mean Change From Baseline to Day 365 in Alanine Aminotransferase, Aspartate Aminotransferase, G-Glutamyl Transferase, and Alkaline Phosphatase
Description: alanine aminotransferase (ALT): >3 x ULN; aspartate aminotransferase (AST): >3 x ULN; G-Glutamyl transferase (GGT): >2 x ULN; Alkaline phosphatase (ALP): >2 x ULN
Time Frame: Baseline (Day 1), Day 365
Population: as for outcome 30
Measure: Mean (Standard Error); unit: U/L
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 131 | 136 | 104
U/L
  ALT (n=131, n=135, n=104) | 3.51 (1.33) | 2.19 (2.31) | -0.04 (1.68)
  AST (n=131, n=135, n=104) | 0.54 (1.04) | -0.11 (1.51) | -2.23 (1.41)
  GGT (n=131, n=135, n=104) | 2.53 (2.81) | -0.61 (1.76) | -2.32 (2.73)
  ALP (n=131, n=136, n=104) | -0.53 (2.16) | -7.78 (2.24) | -4.34 (2.48)

38. Primary Outcome: OL; Mean Change From Baseline to Day 729 in Hemoglobin, Total Protein, and Albumin
Description: Hemoglobin (HGB): >3 g/dL decrease from BL; total protein: < 0.9 x LLN, >1.1 x ULN; albumin:<0.9 x LLN
Time Frame: Baseline (Day 1), Day 729
Population: as for outcome 30
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 124 | 127 | 102
g/dL
  HGB (n=124, n=125, n=102) | 0.66 (0.10) | 0.48 (0.10) | 0.40 (0.13)
  Total protein (n=124, n=127, n=102) | -0.33 (0.05) | -0.25 (0.04) | -0.29 (0.05)
  Albumin (n=124, n=127, n=102) | 0.13 (0.03) | 0.10 (0.03) | 0.06 (0.03)

39. Primary Outcome: OL; Mean Change From Baseline to Day 729 in Platelets
Description: Platelets (PLT): <0.67 x LLN, >1.5 x ULN
Time Frame: Baseline (Day 1), Day 729
Population: as for outcome 30
Measure: Mean (Standard Error); unit: 10^9 c/L
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 124 | 122 | 100
10^9 c/L | -63.9 (6.04) | -5832 (7.66) | -47.7 (8.16)

40. Primary Outcome: OL; Mean Change From Baseline to Day 729 in Hematocrit
Description: Hematocrit: <0.75 x BL
Time Frame: Baseline (Day 1), Day 729
Population: as for outcome 30
Measure: Mean (Standard Error); unit: percentage of red blood cells
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 124 | 124 | 102
percentage of red blood cells | 1.72 (0.29) | 1.23 (0.29) | 0.99 (0.38)

41. Secondary Outcome: OL; Mean Change From Baseline Over Time in DAS 28 (ESR) Score
Description: as for outcome 2
Time Frame: Baseline (Day 1), Day 365, Day 533, Day 729
Population: Number of Participants Analyzed=All Treated Population, all participants who entered the open-label period and received at least one dose of abatacept at any time during this period. Treatment groups represent treatment received in the DB period.n=number of participants with data available.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- ABA + MTX [DB]: Abatacept was administered intravenously (IV) on Days 1, 15, 29 and every 28 days thereafter for a total of 14 doses. Administration was as follows: 500 mg for participants <60 kg, 750 mg for participants 60 to 100 kg and 1 gram for participants >100 kg. All participants received a stable dose of MTX (minimum 15 mg weekly).
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 132 | 136 | 104
units on a scale
  Day 365 (n=122, n=130, n=94) | -3.12 (0.13) | -2.39 (0.13) | -2.81 (0.16)
  Day 533 (n=118, n=121, n=92) | -3.21 (0.13) | -3.04 (0.13) | -2.84 (0.17)
  Day 729 (n=110, n=121, n=93) | -3.35 (0.14) | -3.29 (0.12) | -2.98 (0.17)

42. Secondary Outcome: OL; Percentage of Participants With DAS28 (ESR) Remission and Low Disease Activity (LDAS) Over Time
Description: as for outcome 2
Time Frame: Baseline (Day 1), Day 365, Day 533, Day 729
Population: Number of Participants Analyzed=All Treated Population, all participants who entered the open-label period and received at least one dose of abatacept at any time during this period. Efficacy data was summarized for the 3 DB treatment cohorts.n=number of participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 132 | 136 | 104
percentage of participants
  Day 365 Remission (n=127, n=135, n=102) | 19.7 | 13.3 | 15.7
  Day 365 LDAS (n=127, n=135, n=102) | 37.0 | 23.0 | 29.4
  Day 533 Remission (n=122, n=125, n=98) | 20.5 | 20.0 | 19.4
  Day 533 LDAS (n=122, n=125, n=98) | 37.7 | 33.6 | 35.7
  Day 729 Remission (n=115, n=126, n=100) | 26.1 | 28.6 | 22.0
  Day 729 LDAS (n=115, n=126, n=100) | 41.7 | 45.2 | 34.0

43. Secondary Outcome: OL; Percentage of Participants With Good, Moderate, or No Response According to European League Against Rheumatism (EULAR) Over Time
Description: The DAS28 is a continuous disease measure composite of 4 variables: 28 tender joint count, 28 swollen joint count, ESR or CRP, and participant assessment of disease activity measure on a visual analogue scale. High disease activity= > 5.1, low disease activity= < 3.2, and remission= < 2.6. Clinically significant response= decrease of >1.2 from baseline. Utilizing EULAR response criteria, DAS28 categorical responses define a good (absolute <3.2 or >1.2 improvement from baseline [BL]), moderate (absolute 3.2-5.1 or 0.6-1.2 change from BL), or no response (absolute >5.1 or <0.6 change from BL)
Time Frame: DB Days 365, 533, and 729
Population: as for outcome 41
Measure: Number; unit: percentage of participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 132 | 136 | 104
percentage of participants
  Day 365 Good response (n=122, n=130, n=94) | 38.5 | 23.1 | 30.9
  Day 365 Moderate response (n=122, n=130, n=94) | 53.3 | 58.5 | 55.3
  Day 365 No response (n=122, n=130, n=94) | 8.2 | 18.5 | 13.8
  Day 533 Good response (n=118, n=121, n=92) | 38.1 | 33.1 | 35.9
  Day 533 Moderate response (n=118, n=121, n=92) | 58.5 | 58.7 | 53.3
  Day 533 No response (n=118, n=121, n=92) | 3.4 | 8.3 | 10.9
  Day 729 Good response (n=110, n=121, n=93) | 41.8 | 45.5 | 34.4
  Day 729 Moderate response (n=110, n=121, n=93) | 53.6 | 47.9 | 51.6
  Day 729 No response (n=110, n=121, n=93) | 4.5 | 6.6 | 14.0

44. Secondary Outcome: OL; Percentage of Participants With American College of Rheumatology (ACR) Responses Over Time
Description: as for outcome 11
Time Frame: DB Day 197, Day 365, Day 533, Day 729
Population: as for outcome 30
Measure: Number; unit: percentage of participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 132 | 136 | 104
percentage of participants
  Day 197, ACR 20 (n=130, n=133, n=102) | 73.1 | 68.4 | 44.1
  Day 197, ACR 50 (n=129, n=134, n=103) | 45.7 | 42.5 | 21.4
  Day 197, ACR 70 (n=130, n=133, n=103) | 23.1 | 27.1 | 10.7
  Day 365, ACR 20 (n=130, n=136, n=103) | 88.5 | 69.1 | 75.7
  Day 365, ACR 50 (n=131, n=136, n=102) | 55.0 | 43.4 | 54.9
  Day 365, ACR 70 (n=131, n=136, n=102) | 31.3 | 23.5 | 31.4
  Day 533, ACR 20 (n=128, n=128, n=102) | 82.8 | 82.8 | 74.5
  Day 533, ACR 50 (n=129, n=128, n=103) | 58.1 | 57.0 | 47.6
  Day 533, ACR 70 (n=129, n=127, n=102) | 35.7 | 40.9 | 32.4
  Day 729, ACR 20 (n=119, n=127, n=102) | 86.6 | 84.3 | 76.5
  Day 729, ACR 50 (n=117, n=127, n=101) | 60.7 | 70.9 | 49.5
  Day 729, ACR 70 (n=120, n=127, n=100) | 40.8 | 44.9 | 33.0

45. Secondary Outcome: OL; Percentage of Participants Who Achieved Major Clinical Response
Description: Major Clinical Response was defined as a continuous ACR 70 for six months.
Time Frame: Defined from the date of achieving ACR 70 response to 6 months post response
Population: Protocol-specified analyses of the proportion of participants achieving a Major Clinical Response were not performed since ACR responses in the open-label period could only be assessed at 6-month intervals due to the fact that CRP and ESR were only measured every 6 months during this period.
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 0 | 0 | 0

46. Secondary Outcome: OL; Percentage of Participants With Clinically Meaningful Health Assessment Questionnaire-Disability Index (HAQ-DI) Response Over Time
Description: as for outcome 4
Time Frame: OL Days 197, 253, 281, 309, 337, 365, 449, 533, 617, and 729
Population: as for outcome 41
Measure: Number; unit: percentage of participants
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 132 | 136 | 104
percentage of participants
  Day 197 (n=131, n=134, n=103) | 70.2 | 68.7 | 42.7
  Day 225 (n=132, n=133, n=101) | 75.0 | 72.9 | 52.5
  Day 253 (n=130, n=135, n=102) | 71.5 | 65.2 | 57.8
  Day 281 (n=131, n=135, n=102) | 73.3 | 71.9 | 52.0
  Day 309 (n=131, n=134, n=102) | 71.0 | 70.1 | 62.7
  Day 337 (n=130, n=136, n=101) | 71.5 | 72.1 | 63.4
  Day 365 (n=130, n=136, n=103) | 70.8 | 67.6 | 61.2
  Day 449 (n=129, n=133, n=101) | 70.5 | 72.9 | 64.4
  Day 533 (n=128, n=127, n=103) | 74.2 | 78.0 | 61.2
  Day 617 (n=123, n=127, n=103) | 78.9 | 79.5 | 64.1
  Day 729 (n=122, n=127, n=103) | 74.6 | 78.0 | 63.1

47. Secondary Outcome: OL; Adjusted Mean Change From Baseline to Day 729 in HAQ-DI
Description: as for outcome 4
Time Frame: Day 1 (Baseline), Day 729
Population: All Treated Population, all participants who entered the open-label period and received at least one dose of abatacept at any time during this period. Treatment groups represent treatment received in the DB period.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 122 | 127 | 103
units on a scale
  HAQ-DI | -0.83 (0.06) | -0.84 (0.06) | -0.64 (0.07)
  HAQ-DI component: dressing and grooming | -0.93 (0.08) | -91.0 (0.08) | -0.68 (0.09)
  HAQ-DI component: arising | -0.8 (0.09) | -0.77 (0.08) | -0.72 (0.09)
  HAQ-DI component: eating | -0.86 (0.09) | -0.99 (0.09) | -0.82 (0.10)
  HAQ-DI component: walking | -0.78 (0.09) | -0.73 (0.08) | -0.54 (0.08)
  HAQ-DI component: hygiene | -0.65 (0.10) | -0.65 (0.08) | -0.5 (0.09)
  HAQ-DI component: reach | -0.97 (0.09) | -0.94 (0.10) | -0.64 (0.09)
  HAQ-DI component: grip | -0.88 (0.09) | -0.96 (0.09) | -0.61 (0.09)
  HAQ-DI component: activities | -0.75 (0.09) | -0.73 (0.09) | -0.61 (0.09)

48. Primary Outcome: OL; Mean Change From Baseline to Day 729 in White Blood Cells
Description: as for outcome 33
Time Frame: Baseline (Day 1), Day 729
Population: as for outcome 30
Measure: Mean (Standard Error); unit: 10^3 c/uL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 124 | 125 | 102
10^3 c/uL
  Leukocytes (n=124, n=125, n=102) | -1.57 (0.23) | -1.23 (0.26) | -1.28 (0.23)
  Neutrophils + bands (n=123, n=123, n=101) | -1.62 (0.21) | -1.35 (0.23) | -1.33 (0.22)
  Basophils (n=123, n=123, n=101) | -0.01 (0.00) | 0.00 (0.00) | -0.01 (0.00)
  Monocytes (n=123, n=123, n=101) | -0.05 (0.02) | -0.02 (0.04) | -0.03 (0.02)
  Eosinophils (n=123, n=123, n=101) | -0.01 (0.01) | -0.03 (0.02) | -0.05 (0.02)
  Lymphocytes (n=123, n=123, n=101) | 0.13 (0.06) | 0.18 (0.06) | 0.08 (0.06)

49. Primary Outcome: OL; Mean Change From Baseline to Day 729 in Erythrocytes
Description: Erythrocytes: <0.75 x BL
Time Frame: Baseline (Day 1), Day 729
Population: as for outcome 30
Measure: Mean (Standard Error); unit: 10^6 c/uL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 124 | 125 | 102
10^6 c/uL | 0.07 (0.03) | 0.04 (0.03) | 0.02 (0.04)

50. Primary Outcome: OL; Mean Change From Baseline to Day 729 in Electrolytes
Description: Sodium (Na): <0.95 x LLN, >1.05 x ULN; potassium (K): <0.9 x LLN, >1.1 x ULN; chloride (Cl): <0.9 x LLN, >1.1 x ULN
Time Frame: Baseline (Day 1), Day 729
Population: as for outcome 30
Measure: Mean (Standard Error); unit: mEq/L
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 124 | 127 | 102
mEq/L
  Na | -1.10 (0.28) | -1.12 (0.29) | -1.22 (0.38)
  K | -0.03 (0.04) | -0.04 (0.04) | -0.02 (0.04)
  Cl | -1.31 (0.26) | -1.28 (0.31) | -2.03 (0.29)

51. Primary Outcome: OL; Mean Change From Baseline to Day 729 in Bilirubin, Blood Urea Nitrogen, Creatinine, Calcium, Phosphorous, Serum Glucose, Fasting Serum Glucose, and Uric Acid
Description: as for outcome 36
Time Frame: Baseline (Day 1), Day 729
Population: as for outcome 30
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 124 | 127 | 102
mg/dL
  Creatinine (n=124, n=127, n=102) | 0.08 (0.02) | 0.08 (0.01) | 0.07 (0.02)
  BUN (n=124, n=127, n=102) | -0.37 (0.43) | -0.12 (0.44) | 0.20 (0.46)
  Ca (n=124, n=127, n=102) | 0.01 (0.04) | -0.01 (0.05) | 0.02 (0.05)
  P (n=124, n=127, n=102) | -0.05 (0.05) | -0.16 (0.06) | -0.08 (0.06)
  Uric Acid (n=124, n=127, n=102) | -0.22 (0.08) | -0.02 (0.09) | -0.10 (0.12)
  Total bilirubin (n=124, n=127, n=101) | 0.01 (0.02) | 0.04 (0.02) | 0.03 (0.02)
  Serum glucose (n=123, n=126, n=101) | 9.92 (3.04) | 7.52 (2.02) | 3.74 (2.17)

52. Primary Outcome: OL; Mean Change From Baseline to Day 729 in Alanine Aminotransferase, Aspartate Aminotransferase, G-Glutamyl Transferase, and Alkaline Phosphatase
Description: as for outcome 37
Time Frame: Baseline (Day 1), Day 729
Population: as for outcome 30
Measure: Mean (Standard Error); unit: U/L
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 124 | 127 | 102
U/L
  ALT | 2.73 (1.59) | 1.02 (1.83) | -0.89 (1.96)
  AST | 0.03 (1.17) | -0.22 (1.22) | -2.45 (1.60)
  GGT | 1.23 (2.38) | -0.41 (2.14) | -1.93 (2.95)
  ALP | -0.55 (2.17) | -2.61 (2.83) | -3.91 (3.41)

53. Primary Outcome: OL; Mean Change From Baseline to Day 1121 in Hemoglobin, Total Protein, and Albumin
Description: Hemoglobin (HGB): >3 g/dL decrease from BL; total protein: < 0.9 x LLN, >1.1 x ULN; albumin:<0.9 x LLN
Time Frame: Baseline (Day 1), Day 1121
Population: as for outcome 30
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 102 | 98 | 86
g/dL
  HGB (n=102, n=98, n=85) | 0.66 (0.13) | 0.53 (0.14) | 0.57 (0.13)
  Total protein (n=102, n=98, n=86) | -0.35 (0.05) | -0.24 (0.05) | -0.33 (0.05)
  Albumin (n=102, n=98, n=86) | 0.04 (0.04) | 0.08 (0.04) | -0.01 (0.04)

54. Primary Outcome: OL; Mean Change From Baseline to Day 1121 in Platelets
Description: Platelets (PLT): <0.67 x LLN, >1.5 x ULN
Time Frame: Baseline (Day 1), Day 1121
Population: as for outcome 30
Measure: Mean (Standard Error); unit: 10^9 c/L
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 101 | 95 | 85
10^9 c/L | -67.5 (7.49) | -66.1 (8.86) | -62.5 (8.05)

55. Primary Outcome: OL; Mean Change From Baseline to Day 1121 in Hematocrit
Description: Hematocrit: <0.75 x BL
Time Frame: Baseline (Day 1), Day 1121
Population: as for outcome 30
Measure: Mean (Standard Error); unit: percentage of red blood cells
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 100 | 98 | 85
percentage of red blood cells | 1.83 (0.37) | 1.50 (0.39) | 1.47 (0.39)

56. Primary Outcome: OL; Mean Change From Baseline to Day 1121 in White Blood Cells
Description: as for outcome 33
Time Frame: Baseline (Day 1), Day 1121
Population: as for outcome 30
Measure: Mean (Standard Error); unit: 10^3 c/uL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 102 | 98 | 85
10^3 c/uL
  Leukocytes (n=102, n=98, n=85) | -1.07 (0.27) | -1.09 (0.26) | -0.99 (0.25)
  Neutrophils + bands (n=99, n=96, n=84) | -1.17 (0.25) | -1.40 (0.25) | -1.28 (0.24)
  Basophils (n=99, n=96, n=85) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Monocytes (n=99, n=96, n=84) | 0.03 (0.02) | 0.00 (0.03) | 0.01 (0.03)
  Eosinophils (n=99, n=96, n=84) | 0.00 (0.01) | -0.06 (0.02) | -0.04 (0.02)
  Lymphocytes (n=99, n=96, n=84) | 0.16 (0.08) | 0.34 (0.07) | 0.32 (0.10)

57. Primary Outcome: OL; Mean Change From Baseline to Day 1121 in Erythrocytes
Description: Erythrocytes: <0.75 x BL
Time Frame: Baseline (Day 1), Day 1121
Population: as for outcome 30
Measure: Mean (Standard Error); unit: 10^6 c/uL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 102 | 98 | 85
10^6 c/uL | 0.11 (0.03) | 0.11 (0.04) | 0.12 (0.04)

58. Primary Outcome: OL; Mean Change From Baseline to Day 1121 in Electrolytes
Description: Sodium (Na): <0.95 x LLN, >1.05 x ULN; potassium (K): <0.9 x LLN, >1.1 x ULN; chloride (Cl): <0.9 x LLN, >1.1 x ULN
Time Frame: Baseline (Day 1), Day 1121
Population: as for outcome 30
Measure: Mean (Standard Error); unit: mEq/L
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 102 | 98 | 86
mEq/L
  Na (n=102, n=98, n=86) | -1.80 (0.33) | -1.38 (0.38) | -1.34 (0.42)
  K (n=102, n=98, n=85) | 0.01 (0.04) | 0.08 (0.05) | 0.01 (0.05)
  Cl (n=102, n=98, n=86) | -0.88 (0.35) | -0.94 (0.38) | -1.42 (0.37)

59. Primary Outcome: OL; Mean Change From Baseline to Day 1121 in Bilirubin, Blood Urea Nitrogen, Creatinine, Calcium, Phosphorous, Serum Glucose, Fasting Serum Glucose, and Uric Acid
Description: as for outcome 36
Time Frame: Baseline (Day 1), Day 1121
Population: as for outcome 30
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 102 | 98 | 86
mg/dL
  Creatinine (n=102, n=98, n=86) | 0.06 (0.02) | 0.07 (0.03) | 0.08 (0.02)
  BUN (n=102, n=98, n=86) | -0.04 (0.49) | 0.34 (0.73) | 0.20 (0.56)
  Ca (n=102, n=98, n=86) | -0.01 (0.05) | -0.03 (0.06) | 0.04 (0.05)
  P (n=102, n=98, n=85) | -0.18 (0.07) | -0.19 (0.07) | -0.11 (0.06)
  Uric Acid (n=102, n=98, n=86) | -0.05 (0.11) | 0.13 (0.10) | 0.20 (0.15)
  Total bilirubin (n=102, n=98, n=86) | 0.02 (0.02) | 0.03 (0.02) | 0.03 (0.02)
  Serum glucose (n=101, n=98, n=85) | 12.99 (3.31) | 6.91 (2.10) | 9.07 (3.20)

60. Primary Outcome: OL; Mean Change From Baseline to Day 1121 in Alanine Aminotransferase, Aspartate Aminotransferase, G-Glutamyl Transferase, and Alkaline Phosphatase
Description: as for outcome 37
Time Frame: Baseline (Day 1), Day 1121
Population: as for outcome 30
Measure: Mean (Standard Error); unit: U/L
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 102 | 98 | 86
U/L
  ALT (n=102, n=98, n=86) | 4.74 (1.95) | 4.66 (2.88) | -0.35 (2.33)
  AST (n=102, n=98, n=86) | 3.79 (1.60) | 4.49 (2.13) | 0.38 (1.69)
  GGT (n=102, n=98, n=86) | 1.60 (2.79) | -2.88 (2.16) | -0.14 (3.79)
  ALP (n=88, n=79, n=69) | 1.25 (2.62) | -4.03 (3.79) | -7.35 (3.53)

61. Primary Outcome: OL; Mean Change From Baseline to Day 1513 in Hemoglobin, Total Protein, and Albumin
Description: Hemoglobin (HGB): >3 g/dL decrease from BL; total protein: < 0.9 x LLN, >1.1 x ULN; albumin:<0.9 x LLN
Time Frame: Baseline (Day 1), Day 1513
Population: as for outcome 30
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 23 | 20 | 16
g/dL
  HGB | 0.25 (0.33) | 0.44 (0.31) | 0.56 (0.32)
  Total protein | -0.73 (0.09) | -0.33 (0.11) | -0.34 (0.14)
  Albumin | -0.06 (0.07) | 0.10 (0.07) | 0.00 (0.11)

62. Primary Outcome: OL; Mean Change From Baseline to Day 1513 in Platelets
Description: Platelets (PLT): <0.67 x LLN, >1.5 x ULN
Time Frame: Baseline (Day 1), Day 1513
Population: as for outcome 30
Measure: Mean (Standard Error); unit: 10^9 c/L
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 23 | 19 | 16
10^9 c/L | -78.0 (17.20) | -74.0 (16.18) | -99.2 (19.83)

63. Primary Outcome: OL; Mean Change From Baseline to Day 1513 in Hematocrit
Description: Hematocrit: <0.75 x BL
Time Frame: Baseline (Day 1), Day 1513
Population: as for outcome 30
Measure: Mean (Standard Error); unit: percentage of red blood cells
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 23 | 19 | 16
percentage of red blood cells | 0.92 (1.00) | 1.28 (0.92) | 1.18 (1.00)

64. Primary Outcome: OL; Mean Change From Baseline to Day 1513 in White Blood Cells
Description: as for outcome 33
Time Frame: Baseline (Day 1), Day 1513
Population: as for outcome 30
Measure: Mean (Standard Error); unit: 10^3 c/uL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 23 | 20 | 16
10^3 c/uL
  Leukocytes (n=23, n=20, n=16) | -0.34 (0.45) | -1.08 (0.63) | -2.13 (0.50)
  Neutrophils + bands (n=22, n=17, n=16) | -0.37 (0.33) | -1.03 (0.68) | -1.93 (0.50)
  Basophils (n=22, n=17, n=16) | 0.00 (0.01) | -0.01 (0.01) | -0.01 (0.01)
  Monocytes (n=22, n=17, n=16) | 0.01 (0.03) | -0.10 (0.09) | -0.05 (0.04)
  Eosinophils (n=22, n=17, n=16) | 0.04 (0.06) | -0.11 (0.16) | -0.23 (0.00)
  Lymphocytes (n=22, n=17, n=16) | 0.20 (0.14) | 0.16 (0.16) | -0.15 (0.16)

65. Primary Outcome: OL; Mean Change From Baseline to Day 1513 in Erythrocytes
Description: Erythrocytes: <0.75 x BL
Time Frame: Baseline (Day 1), Day 1513
Population: as for outcome 30
Measure: Mean (Standard Error); unit: 10^6 c/uL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 23 | 19 | 16
10^6 c/uL | -0.10 (0.09) | 0.00 (0.09) | -0.09 (0.08)

66. Primary Outcome: OL; Mean Change From Baseline to Day 1513 in Electrolytes
Description: Sodium (Na): <0.95 x LLN, >1.05 x ULN; potassium (K): <0.9 x LLN, >1.1 x ULN; chloride (Cl): <0.9 x LLN, >1.1 x ULN
Time Frame: Baseline (Day 1), Day 1513
Population: as for outcome 30
Measure: Mean (Standard Error); unit: mEq/L
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 23 | 20 | 16
mEq/L
  Na (n=22, n=20, n=16) | -4.36 (0.73) | -3.80 (0.99) | -4.50 (0.74)
  K (n=23, n=20, n=16) | -0.16 (0.10) | -0.32 (0.08) | -0.46 (0.11)
  Cl (n=23, n=20, n=16) | -2.48 (0.71) | -2.60 (0.84) | -4.13 (0.88)

67. Primary Outcome: OL; Mean Change From Baseline to Day 1513 in Bilirubin, Blood Urea Nitrogen, Creatinine, Calcium, Phosphorous, Serum Glucose, Fasting Serum Glucose, and Uric Acid
Description: as for outcome 36
Time Frame: Baseline (Day 1), Day 1513
Population: as for outcome 30
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 23 | 20 | 16
mg/dL
  Creatinine | 0.10 (0.02) | 0.05 (0.04) | 0.08 (0.06)
  BUN | 2.87 (0.90) | -0.40 (1.13) | 0.63 (1.36)
  Ca | 0.27 (0.07) | 0.38 (0.09) | 0.35 (0.12)
  P | -0.09 (0.11) | -0.51 (0.16) | -0.17 (0.13)
  Uric Acid | 0.03 (0.18) | 0.06 (0.21) | 0.33 (0.33)
  Total bilirubin | 0.08 (0.10) | 0.09 (0.03) | 0.23 (0.14)
  Serum glucose | 8.87 (3.19) | 9.00 (1.88) | 8.44 (4.38)

68. Primary Outcome: OL; Mean Change From Baseline to Day 1513 in Alanine Aminotransferase, Aspartate Aminotransferase, G-Glutamyl Transferase, and Alkaline Phosphatase
Description: as for outcome 37
Time Frame: Baseline (Day 1), Day 1513
Population: as for outcome 30
Measure: Mean (Standard Error); unit: U/L
Arm/Group | ABA + MTX [DB] | INF + MTX [DB] | PLA + MTX [DB]
Number analyzed (Participants) | 23 | 20 | 16
U/L
  ALT | -1.87 (2.73) | -9.20 (3.75) | 2.44 (8.07)
  AST | -1.35 (1.72) | -2.85 (2.55) | 0.38 (7.23)
  GGT | -3.00 (2.99) | -10.9 (5.79) | -3.06 (10.30)
  ALP | -15.8 (5.23) | -18.7 (7.12) | -11.30 (7.80)

69. Primary Outcome: OL; Mean Systolic (SBP) and Diastolic (DBP) Blood Pressure During Open Label Period
Description: Seated Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP), units=mm mercury (Hg)
Time Frame: Days 365, 729, 1121, and 1513
Population: Number of Participants Analyzed=All Treated Population, all participants who entered the open-label period and received at least one dose of abatacept at any time during this period.n=number of participants with data available.
Measure: Mean (Standard Deviation); unit: mm mercury (Hg)
Arm/Group | ABA + MTX [OL]
Number analyzed (Participants) | 372
mm mercury (Hg)
  Day 365 SBP pre-dose (n=343) | 119.0 (15.03)
  Day 365 SBP post-dose (n=341) | 118.8 (15.35)
  Day 729 SBP pre-dose (n=321) | 120.4 (15.20)
  Day 729 SBP post-dose (n=323) | 119.5 (15.02)
  Day 1121 SBP pre-dose (n=265) | 121.1 (15.59)
  Day 1121 SBP post-dose (n=265) | 119.2 (13.99)
  Day 1513 SBP pre-dose (n=52) | 114.6 (13.57)
  Day 1513 SBP post-dose (n=52) | 114.2 (12.90)
  Day 365 DBP pre-dose (n=343) | 74.5 (9.80)
  Day 365 DBP post-dose (n=341) | 74.0 (10.18)
  Day 729 DBP pre-dose (n=321) | 74.9 (9.69)
  Day 729 DBP post-dose (n=323) | 74.6 (9.92)
  Day 1121 DBP pre-dose (n=265) | 74.9 (9.45)
  Day 1121 DBP post-dose (n=265) | 73.6 (9.12)
  Day 1513 DBP pre-dose (n=52) | 71.7 (9.45)
  Day 1513 DBP post-dose (n=52) | 72.1 (9.11)

70. Primary Outcome: OL; Mean Heart Rate (HR) During Open Label Period
Description: Heart Rate (HR), units=beats per minute (bpm)
Time Frame: Days 365, 729, 1121, and 1513
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | ABA + MTX [OL]
Number analyzed (Participants) | 372
beats per minute (bpm)
  Day 365 HR pre-dose (n=343) | 74.2 (9.30)
  Day 365 HR post-dose (n=341) | 74.1 (8.57)
  Day 729 HR pre-dose (n=322) | 74.2 (9.12)
  Day 729 HR post-dose (n=324) | 73.4 (8.59)
  Day 1121 HR pre-dose (n=265) | 73.9 (9.31)
  Day 1121 HR post-dose (n=265) | 73.8 (9.46)
  Day 1513 HR pre-dose (n=52) | 73.0 (8.38)
  Day 1513 HR post-dose (n=52) | 73.8 (7.16)

71. Primary Outcome: OL; Mean Temperature (T) During Open Label Period
Description: Temperature (T), units=degrees Celcius
Time Frame: Days 365, 729, 1121, and 1513
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | ABA + MTX [OL]
Number analyzed (Participants) | 372
degrees Celsius
  Day 365 T pre-dose (n=339) | 36.3 (0.43)
  Day 365 T post-dose (n=339) | 36.3 (0.41)
  Day 729 T pre-dose (n=320) | 36.3 (0.45)
  Day 729 T post-dose (n=323) | 36.3 (0.42)
  Day 1121 T pre-dose (n=263) | 36.2 (0.51)
  Day 1121 T post-dose (n=264) | 36.2 (0.47)
  Day 1513 T pre-dose (n=52) | 36.1 (0.35)
  Day 1513 T post-dose (n=52) | 36.1 (0.37)

ADVERSE EVENTS:
Groups:
- ABA (DB): Abatacept was administered intravenously (IV) on Days 1, 15, 29 and every 28 days thereafter for a total of 14 doses. Administration was as follows: 500 mg for participants < 60 kg, 750 mg for participants 60 to 100 kg and 1 gram for participants > 100 kg. All participants received a stable dose of MTX (minimum 15 mg weekly).
- PLA + MTX [DB]: Normal saline was administered as placebo. All participants received a stable dose of MTX (minimum 15 mg weekly). After placebo treatment from Day 1-197, 104 participants were reallocated to receive abatacept (weight based) plus a stable dose of MTX (minimum 15 mg weekly).
Arm/Group | ABA (DB) | ABA + MTX [OL] | INF + MTX [DB] | PLA + MTX [DB]
Serious Adverse Events (participants affected / at risk) | 17/156 | 90/372 | 30/165 | 21/110
Other Adverse Events (participants affected / at risk) | 105/156 | 285/372 | 130/165 | 82/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABA (DB) (N=156) | ABA + MTX [OL] (N=372) | INF + MTX [DB] (N=165) | PLA + MTX [DB] (N=110)
CATARACT (Eye disorders) | 0 | 1 | 0 | 0
CORNEAL PERFORATION (Eye disorders) | 0 | 1 | 0 | 0
HORMONE LEVEL ABNORMAL (Investigations) | 0 | 1 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 1
ARRHYTHMIA (Cardiac disorders) | 0 | 1 | 0 | 0
PERICARDITIS (Cardiac disorders) | 0 | 0 | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 1 | 1 | 1 | 0
ANGINA UNSTABLE (Cardiac disorders) | 1 | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 1 | 1 | 0
ATRIAL TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 3 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 1 | 0 | 0
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 1 | 0 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 2 | 0 | 0
ARTERITIS (Vascular disorders) | 0 | 0 | 1 | 0
HAEMATOMA (Vascular disorders) | 0 | 0 | 1 | 0
VASCULITIS (Vascular disorders) | 1 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 1 | 0
AORTIC STENOSIS (Vascular disorders) | 0 | 1 | 0 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 0 | 0 | 0
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1 | 0 | 0
BILIARY COLIC (Hepatobiliary disorders) | 0 | 0 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 2 | 1 | 0
ANAPHYLACTIC SHOCK (Immune system disorders) | 0 | 0 | 0 | 1
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
ANAL FISSURE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ANAL SKIN TAGS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
HYPERTROPHIC ANAL PAPILLA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
SEPSIS (Infections and infestations) | 0 | 0 | 0 | 1
ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 2 | 1 | 3 | 1
SINUSITIS (Infections and infestations) | 1 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 3 | 1 | 0
ERYSIPELAS (Infections and infestations) | 0 | 1 | 1 | 0
APPENDICITIS (Infections and infestations) | 0 | 2 | 0 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 0 | 1 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 0 | 1 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1 | 0
LOBAR PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 0
WOUND INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
BURSITIS INFECTIVE (Infections and infestations) | 0 | 0 | 0 | 1
ABSCESS SOFT TISSUE (Infections and infestations) | 0 | 0 | 0 | 1
ENCEPHALITIS HERPES (Infections and infestations) | 0 | 0 | 1 | 0
INFECTED SKIN ULCER (Infections and infestations) | 1 | 0 | 0 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0
NECROTISING FASCIITIS (Infections and infestations) | 0 | 1 | 0 | 0
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 | 0 | 1 | 0
APPENDICITIS PERFORATED (Infections and infestations) | 0 | 0 | 1 | 0
PERITONEAL TUBERCULOSIS (Infections and infestations) | 0 | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 5 | 0 | 0
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 0 | 0 | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 0 | 1 | 1
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 1
BLADDER PROLAPSE (Renal and urinary disorders) | 0 | 1 | 0 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 0 | 0 | 1
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 2 | 0 | 0
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
UTERINE POLYP (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
OVARIAN TORSION (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
UTERINE PROLAPSE (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
ACCIDENT (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
ILIUM FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
CARTILAGE INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
FAILURE OF IMPLANT (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
PUBIC RAMI FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
COMPLICATED FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
DISLOCATION OF JOINT PROSTHESIS (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
FISTULA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 2
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 19 | 4 | 4
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
LARYNGEAL GRANULOMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
PYREXIA (General disorders) | 1 | 2 | 0 | 0
HYPERTHERMIA (General disorders) | 0 | 1 | 0 | 0
LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
FIBROSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
BENIGN LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
MALIGNANT ANORECTAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
BENIGN NEOPLASM OF THYROID GLAND (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABA (DB) (N=156) | ABA + MTX [OL] (N=372) | INF + MTX [DB] (N=165) | PLA + MTX [DB] (N=110)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 6 | 9 | 4 | 6
HYPERTENSION (Vascular disorders) | 13 | 42 | 11 | 13
ANXIETY (Psychiatric disorders) | 5 | 24 | 7 | 2
INSOMNIA (Psychiatric disorders) | 5 | 15 | 12 | 3
DEPRESSION (Psychiatric disorders) | 6 | 26 | 6 | 1
HEADACHE (Nervous system disorders) | 23 | 54 | 34 | 24
DIZZINESS (Nervous system disorders) | 11 | 25 | 13 | 7
NAUSEA (Gastrointestinal disorders) | 16 | 26 | 21 | 10
VOMITING (Gastrointestinal disorders) | 5 | 13 | 10 | 5
DIARRHOEA (Gastrointestinal disorders) | 21 | 56 | 21 | 7
DYSPEPSIA (Gastrointestinal disorders) | 19 | 41 | 17 | 7
GASTRITIS (Gastrointestinal disorders) | 6 | 22 | 8 | 7
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 23 | 8 | 2
INFLUENZA (Infections and infestations) | 13 | 49 | 12 | 6
SINUSITIS (Infections and infestations) | 10 | 29 | 7 | 8
BRONCHITIS (Infections and infestations) | 11 | 41 | 10 | 11
PHARYNGITIS (Infections and infestations) | 12 | 43 | 17 | 9
GASTROENTERITIS (Infections and infestations) | 4 | 23 | 12 | 6
NASOPHARYNGITIS (Infections and infestations) | 20 | 69 | 26 | 15
URINARY TRACT INFECTION (Infections and infestations) | 8 | 67 | 18 | 13
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 | 50 | 19 | 16
RASH (Skin and subcutaneous tissue disorders) | 1 | 12 | 10 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 5 | 5 | 10 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 3 | 10 | 11 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 12 | 41 | 10 | 8
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 28 | 7 | 5
OEDEMA PERIPHERAL (General disorders) | 8 | 18 | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.